CLINICAL TRIAL: NCT04733794
Title: Feasibility of Implementing a Comprehensive, Patient-Centered Approach to Bowel Dysfunction After Low Anterior Resection for Rectal Cancer
Brief Title: Feasibility Bowel Dysfunction Program After Low Anterior Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-8016
Record Dates: First submitted 2017-10-30; First posted 2021-02-02 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Rectal Cancer; Low Anterior Resection
Keywords: Bowel Dysfunction; Low Anterior Resection; Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms; Intestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgery for Stoma Reversal (Experimental): All study participants will receive stoma reversal, complete baseline questionnaire, pelvic floor training and follow up questionnaires
  Interventions: Procedure: Stoma reversal

INTERVENTIONS:
Procedure: Stoma reversal — Patients will receive a comprehensive intervention to addresses bowel, sexual, and urinary dysfunction. Patients meeting appropriate inclusion criteria will be approached at a clinic visit with their surgeon. If they agree to participate, they will complete an initial baseline questionnaire. Questionnaires will be distributed on iPads during their clinic visit

SUMMARY:
This study will facilitate a better understanding of the overall experience of our rectal cancer survivors after Low Anterior Resection for rectal cancer. Studies have demonstrated that the development of bowel and genitourinary dysfunction after this procedure is very distressing to patients and can have a significant impact on overall quality of life. By providing interventions that can be performed at home, investigator may alleviate these symptoms in hopes of improving the experience of patients undergoing Low Anterior Resection. By acknowledging these potentially debilitating symptoms in a systematic way, the investigator hopes to reinforce the importance of symptom management in the survivorship phase after treatment has been completed and ultimately facilitate an individual's return to routine activities.

DETAILED DESCRIPTION:
Subjects will be recruited from patients presenting to the surgical oncology clinic at Fox Chase Cancer Center. These patients will have already undergone Low Anterior Resection with a diverting stoma (colostomy or ileostomy) and will be planning on undergoing reversal of their stoma in the near future. Subjects will be recruited over a period of 1 year. Such clinic patients' medical records will be reviewed to determine whether they are possible candidates for inclusion in the study. They will be identified based on their diagnosis of either Stage II or III rectal cancer as stated in prior clinic notes, pathology reports, or radiologic image reports. Participants must have previously undergone Low Anterior Resection with a diverting stoma and the surgical plan must be for them to undergo ostomy reversal. They will be approached during a clinic visit by either a co-investigator or a member of the surgery team (fellow or surgeon) or a research coordinator delegate and asked to participate in the research study. They will be given a document for informed consent that will describe the study and potential risks and benefits to the patient. The investigators plan to enroll 10 patients at Fox Chase Cancer Center. Subjects will receive no monetary compensation

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Stage II or III rectal cancer, a history of having an LAR with diverting stoma, and a plan to undergo stoma reversal within the next 6 months

Exclusion Criteria:

* Patients enrolled who develop an anastomotic leak at the time of stoma reversal that would necessitate another temporary or permanent stoma, they will be considered unevaluable and will be excluded from the analysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Bowel dysfunction | 12 months
  Symptoms will be assessed at scheduled visits with patient's provider by means of the follow up questionnaire containing 11 questions scored on a scale from 0 to 4 with a minimum score of 1 and a maximum score of 44
Urinary function | 12 months
  Symptoms will be assessed at scheduled visits with patient's provider by means of the follow up questionnaire containing 11 questions scored on a scale from 0 to 4 with a minimum score of 1 and a maximum score of 44
Sexual function | 12 months
  Symptoms will be assessed at scheduled visits with patient's provider by means of the follow up questionnaire containing 8-10 questions (8 for women and 10 for men) scored on a scale from 0 to 4 with a minimum score of 0 and maximum score of 40

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No